CLINICAL TRIAL: NCT04717596
Title: Implementation and Examination of Contraception Care for Hospitalized Adolescents With Mental Health Disorders
Status: Completed | Type: Observational
Sponsor: Elise Berlan (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Elise Berlan, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00001603
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Contraception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: BC4Teens Care — Healthcare providers will be trained in contraceptive counseling and provision.

SUMMARY:
This study is a hybrid trial that examines both the clinical effectiveness and the implementation of BC4Teens Contraception Care. The investigators use a naturalistic one-group longitudinal study design to maximize feasibility and external validity, which is important for understanding implementation and effectiveness in real-world service delivery settings.

DETAILED DESCRIPTION:
Approximately one in five American youth have experienced severe impairment due to mental health disorders, with anxiety and mood disorders being most common among female adolescents. Mental health disorders are associated with a range of sexual risk behaviors and unintended pregnancy. Youth with mental health disorders have higher rates of condom and contraception non-use (especially short acting), earlier sexual debut, and higher fertility rates.

Avoiding an unwanted or unintended pregnancy is particularly important for women with underlying mental health disorders. Experiencing a pregnancy exacerbates underlying mental health disorders in women with mental health disorder. And children born out of an unintended pregnancy or in context of mother with active mental health disorder face additional risks to their wellbeing. Long acting reversible contraceptives (LARCs), i.e. contraceptive implants and intrauterine devices, have attributes that may be particularly attractive to adolescents with mental health disorders. In particular, they are highly effective and do not require ongoing maintenance. However, adolescents with mental health disorders face multiple barriers to accessing contraception care. Novel solutions are needed to improve access to contraception care, including LARC, for adolescents with mental disorders.

The inpatient pediatric hospitalization setting is a missed opportunity for improving adolescent sexual and reproductive health. Nearly 10% of pediatric hospitalizations are for a primary mental health diagnosis, and mood disorders are the most common primary mental health diagnosis among these hospitalizations. Sexual and reproductive healthcare is rarely provided to hospitalized adolescents. At Nationwide Children's Hospital, a chart audit completed in December 2019 found that no adolescents hospitalized for mental health disorders on the Hospital Pediatrics service had documentation they were screened for sexual activity.

Adolescents are interested in learning about sexual and reproductive health and receiving sexual and reproductive healthcare in the hospital setting regardless of age, gender, and prior sexual experiences. Two studies of pediatric hospitalists found that the majority of those physicians felt that sexual and reproductive services are appropriate for hospitalized adolescents, with high support for referrals and starting contraception in the hospital. Numerous barriers to inpatient provision of contraceptives/sexual reproductive healthcare were endorsed, including: concerns about follow up after discharge, lack of knowledge about confidentiality, lack of knowledge about contraception, interference with the treatment plan, time constraints, and pregnancy risk in lesbian, gay, bisexual, and transgender youth. Riese et al. conducted a trial of an interactive patient-facing electronic sexual health module and found that it was acceptable to adolescents and their parents, and that most participants requested a sexual health service after completing the module. (The most requested service was viewing a contraception video made by this PI.) There are no published studies of interventions to improve contraception care to hospitalized adolescents with mental health disorders.

The PI designed an adolescent-friendly contraceptive counseling training course, called BC4Teens Counseling, in use since 2014 by outpatient family planning clinicians in BC4Teens Clinic at Nationwide Children's Hospital, the second largest children's hospital in the US. BC4Teens Counseling is adapted from Contraceptive Choice Project materials and employs efficacy-based counseling, which is endorsed by WHO and American Academy of Pediatrics. This training will be adapted to current best practice recommendations, including shared-decision making. The PI, with a multidisciplinary team, has also designed a comprehensive Contraception Clinical Guideline, contraception initiation job aid, and electronic health record order set with decision support for contraception initiation. These are currently used in outpatient care across several departments at Nationwide Children's Hospital. The PI is a Nexplanon Clinical Trainer and has extensive experience with clinical teaching on contraception care and Nexplanon procedures, and this site is a Merck Center of Experience.

The investigators propose the following BC4Teens Contraception Care Intervention. All healthcare professionals participating the intervention will receive training in the following:

* BC4Teens Counseling is a set of adolescent-friendly contraception counseling and provision protocols for all FDA-approved prescription contraceptives. The training includes up-to-date information about maintaining adolescent confidentiality, coding, and care for sexually transmitted infections.
* Nationwide Children's Contraception Clinical Guideline, a contraception initiation job aid, and electronic health record order set and decision support for contraception initiation. These materials are evidence-based and reference established best practices for contraception care, pregnancy options counseling, and preconception care.
* Nexplanon Clinical Training and credentialing in Nexplanon procedures during planning phase.
* Information about institutional policies, adolescent confidentiality and consent, and local sexual health resources will be provided to participating healthcare professionals.
* Ongoing technical and procedural support from institutional BC4Teens expert trainer.

More than 2000 female adolescents with mental health disorders were hospitalized in 2019 at Nationwide Children's Hospital. In February 2020 The Big Lots Behavioral Health Pavilion (BHP) at Nationwide Children's Hospital opened its doors. The BHP is America's largest center dedicated exclusively to child and adolescent behavioral and mental health on a pediatric medical campus. Due to the impact of COVID and the simultaneous opening of the BHP, adolescents with mental health disorders are now hospitalized differently within the Nationwide Children's Hospital system than before. Presently at Nationwide Children's Hospital adolescents with mental health disorders are admitted to the Psychiatry Unit, the observation unit of the psychiatric crisis department, or the Youth Crisis Stabilization Unit (YCSU). The investigators anticipate that once the initial COVID impact has passed, adolescent patients with mental health disorders may overflow onto the Hospital Pediatrics service within the main hospital as they previously did.

The primary goal of this study is to examine an intervention to improve access to contraception care among female adolescents hospitalized with mental health disorders within Nationwide Children's Hospital.

One of the investigators' long term goals is to scale-up effective contraceptive counseling interventions like BC4Teens Contraception Care beyond Nationwide Children's Hospital to other inpatient settings. This type of scale up has potential to expand the reach of contraceptive care to a broader population of adolescent females with mental health concerns. However, evidence-based psychosocial interventions sometimes fail to yield the same benefits observed in controlled studies when they are transported to new settings. Limited resources, poor alignment with organizational structures and missions, concerns about the interventions' acceptability, and heterogeneity of patient needs and professional skill can lead to difficulty delivering the intervention with fidelity (as it was intended with all core components and at prescribed dosage). This "voltage drop" in intervention effectiveness as it moves into routine care is often attributed to failure to optimize the intervention in its new context.

In this study, the secondary goal is to examine the strategies and processes used to implement BC4Teens at Nationwide Children's Hospital, and create an implementation manual that can be used to scale up this intervention in other settings. Thus, the investigators are embedding a naturalistic observational study of BC4Teens implementation within the effectiveness research. This study component will focus on specifying the procedures used to tailor the intervention and training supports, and monitoring the outcomes of implementation (including the degree to which professionals adopt BC4Teens, deliver it with fidelity, and reach the target population). In addition to informing an implementation manual, these results will also advance understanding of the model including the degree to which the model must be delivered as intended in order to generate clinical benefit, identify types of professionals best suited for delivering BC4Teens, and patients for whom this intervention is considered acceptable.

ELIGIBILITY:
Inclusion Criteria:

* female adolescents, ages 14 and up, receiving care in Psychiatric Unit, Youth Crisis Stabilization Unit (YCSU), Psychiatric Crisis Department Extended Observation Care Unit, and Hospital Pediatrics service

Exclusion Criteria:

* unable to consent due to mental health disorder, serious medical condition, non-English speaking, known pregnancy

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: female adolescents hospitalized for mental health disorder on Psychiatric Unit, Youth Crisis Stabilization Unit (YCSU), Psychiatric Crisis Department Extended Observation Care Unit, and Hospital Pediatrics service at Nationwide Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise Berlan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside of the research team.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort: Single cohort
Period: Overall Study
Arm/Group | Cohort
Started | 455
Completed | 451
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Female adolescents 14 years and older hospitalized for mental health disorders at Nationwide Children's Hospital.
Groups:
- Baseline Cohort: Female adolescents 14 years and older hospitalized for mental health disorders at Nationwide Children's Hospital.
Arm/Group | Baseline Cohort
Number analyzed (Participants) | 451
Age, Continuous [Mean (Full Range); unit: years] | 16.1 [14.1 to 18.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 451
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 89
  Race: White or Caucasian | 295
  Race: Other race/multi-race | 64
  Race: Missing | 3

OUTCOME MEASURES:

1. Primary Outcome: Interest BC4Teens Care
Description: % participants who answer yes to the following question "Interest in learning more about contraception during your hospital stay". Investigators will calculate the percentage of participants who answer yes to the Interest in Contraption Initiation question.
Time Frame: Baseline
Population: Female adolescents 14 years and older hospitalized for mental health disorders having completed this question in the survey
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Cohort
Number analyzed (Participants) | 450
Participants | 231

ADVERSE EVENTS:
Time Frame: 1 day
Description: We used the clinicaltrials.gov definition.
Groups:
- Cohort: Female adolescents 14 years and older hospitalized for mental health disorders at Nationwide Children's Hospital.
Arm/Group | Cohort
All-Cause Mortality (participants affected / at risk) | 0/451
Serious Adverse Events (participants affected / at risk) | 0/451
Other Adverse Events (participants affected / at risk) | 0/451

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT04717596/Prot_SAP_000.pdf